CLINICAL TRIAL: NCT00564590
Title: The Effects of Melatonin on GERD Symptoms and Esophageal Acid Exposure
Brief Title: SThe Effects of Melatonin on GERD Symptoms
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 004548
Record Dates: First submitted 2007-11-26; First posted 2007-11-28 (Estimated); Last update posted 2007-11-28 (Estimated); Status verified 2007-11

CONDITIONS: Gastroesophageal Reflux Disease
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Melatonin; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- A (Experimental): Melatonin treatment group
  Interventions: Drug: Melatonin
- B (Active Comparator): Omeprazole 20 mg once a day for 3 months
  Interventions: Other: omeprazole
- C (Experimental): Placebo once a day for 3 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Melatonin — 4 mg of Melatonin once a day for 3 months
  Arms: A
Other: omeprazole — omeprazole 20 mg once a day
  Other Names: Omepradex
  Arms: B
Drug: Placebo — Placebo once a day
  Arms: C

SUMMARY:
We hypothesize that melatonin as compared to PPI and to placebo, improves GERD symptoms by decreasing esophageal acid exposure and esophageal acid sensitivity in GERD. We hypothesize that melatonin as compared to PPI and to placebo reduce the frequency and duration of transient lower esophageal sphincter relaxations (TLESRs). In addition we hypothesize that melatonin as compared to PPI and to placebo improves quality of life and quality of sleep of GERD patients.

DETAILED DESCRIPTION:
Background: Gastroesophageal reflux disease (GERD) is a chronic, persistent and common medical problem. The standard of care for GERD includes chronic administration of acid-suppressive drugs. However, clinical failure in GERD is increasingly reported.

Aim: To determine the efficacy of treatment with melatonin as compared to standard dose proton pump inhibitor (PPI) as compared to placebo in patients with GERD.

Study objectives: [1] To compare the degree of GERD symptoms improvement and esophageal acid sensitivity before and after treatment. [2] To determine the effect of treatment on the % total, upright and supine time pH <4 using 24-hour esophageal pH monitoring. [3] To determine the effect of treatment on frequency and duration of lower esophageal sphincter relaxation. [4] To compare the quality of life and quality of sleep in GERD patients before and after treatment.

Methods: This is a randomized, double blind, parallel groups study of 150 patients with GERD. Patients with classic heartburn symptoms (heartburn and/or regurgitation) and normal upper endoscopy from the gastroenterology department at Rabin Medical Center will be enrolled into the study. At baseline, all enrolled patients will have 24-hour esophageal pH monitoring and a modified acid perfusion test to assess the extent of distal esophageal acid exposure and esophageal acid sensitivity, respectively. Patients will be evaluated by a demographics questionnaire, the GERD Symptom Questionnaire, the Quality of Sleep questionnaire and the SF-36. Baseline urinary excretion of the main melatonin metabolite, 6-sulfatoxymelatonin (6SMT) will be assessed in all subjects at baseline. Patients will be randomized to either melatonin or standard dose PPI or placebo over a period of 4 weeks. In addition patients will fill a diary on a daily basis that documents severity and frequency of GERD-related symptoms. Symptom score (frequency x severity) will be calculated for previous 7 days at baseline and at the end of treatment in all groups. After 4 weeks of treatment, patients will undergo a second 24-hour esophageal pH monitoring, a modified acid perfusion test and will complete the GERD Symptom Questionnaire, the Quality of Sleep Questionnaire and the SF-36.

Implications: This study will determine if melatonin decreases GERD symptoms, acid esophageal exposure and improves quality of life and sleep in patients with GERD. Furthermore, if there will be a significant clinical response to melatonin it will be possible to add this compound to the treatment armamentum of GERD.

ELIGIBILITY:
INCLUSION CRITERIA:

* Ages 18-75.
* Male or female.
* GERD symptoms at least twice a week for the last three months.
* Able to read, understand and complete study questionnaires and diary
* Understand the study procedures and sign written informed consent.
* Able to comply with all study requirements.

EXCLUSION CRITERIA:

* Subjects with erosive esophagitis (EE), Barrett's esophagus (BE) and esophageal stricture or adenocarcinoma on upper endoscopy.
* Subjects with previous upper gastrointestinal surgery.
* Subjects with clinically significant medical conditions (cardiovascular, respiratory, renal, hepatic, hematologic, endocrine, neurologic and psychiatric); examples as follows: liver cirrhosis, severe COPD, severe renal failure, severe heart failure, active malignancy.
* Subjects requiring narcotics (morphine, methadone, etc.).
* Subjects requiring melatonin
* Subjects with diabetes, scleroderma and neuromuscular disorders.
* Lactating or pregnant women.
* Subjects with an unrecognized lifestyle such as shift workers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2008-10; Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
This study will test the efficacy of melatonin (10 mg once a day) as compared to standard dose PPI (omeprazole 20 mg once a day) and placebo on different subjective and objective parameters of 150 patients with GERD. | 3 years

SECONDARY OUTCOMES:
To determine the effect of melatonin versus standard-dose PPI versus placebo on frequency and duration of TLESRs. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ram M Dickman, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Beilinson Hospital, Petah Tikva, Israel

REFERENCES:
- [Background] Pereira Rde S. Regression of gastroesophageal reflux disease symptoms using dietary supplementation with melatonin, vitamins and aminoacids: comparison with omeprazole. J Pineal Res. 2006 Oct;41(3):195-200. doi: 10.1111/j.1600-079X.2006.00359.x. PMID 16948779